CLINICAL TRIAL: NCT07183579
Title: A Retrospective Observational Study of the Effect of Dosing Regimen of Burosumab on Biochemical Control of Serum Phosphate Levels in Patients With X-linked Hypophosphataemia (XLH)
Brief Title: Effective Dosing of Burosumab in XLH
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Sheffield Children's NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 25033; 291899 (Other: IRAS Project ID)
Record Dates: First submitted 2025-07-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: X-linked Hypophosphatemia (XLH)
Keywords: Hypophosphatemia, X-Linked Dominant; Rickets; Burosumab; Monoclonal Antibodies; Alkaline Phosphatase; Parathyroid Hormone; Retrospective Studies; Observational Study; Multicenter Study; Dose-Response Relationship, Drug; Child; Adolescent; Pediatrics; X-Linked Hypophosphatemia (XLH); Metabolic Bone Disease; Crysvita; FGF23 Antibody; Real-World Evidence; Pragmatic Clinical Study; Serum Phosphate; Nephrocalcinosis; Paediatric Endocrinology; Treatment Outcome; Adverse Events; Drug Administration Schedule
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Hypophosphatemia; Rickets; Bone Diseases, Metabolic; Nephrocalcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- XLH: Children and young people with XLH treated with Burosumab

SUMMARY:
X-linked hypophosphataemia (XLH) is a rare, hereditary condition. The genetic defect leads to low blood phosphate levels and vitamin D suppression. Phosphate is required for strong bones and teeth and to store energy in cells. Low phosphate leads to soft bones (rickets). Patients experience bowed legs, short stature, bone pain and dental pain.

Prior to Burosumab, conventional treatment of XLH previously consisted of two medications. On this regimen, patients take oral phosphate supplements 4-6 times a day and an active form of vitamin D daily. This treatment can leave patients with residual symptoms. They report significant disabilities and reduced quality of life.

Burosumab (Crysvita, Kyowa Kirin) is now the standard paediatric treatment for XLH. It is given once a fortnight by injection under the skin. Early studies used a starting dose of 0.4mg/kg per dose. NICE recommends a starting dose of 0.4mg/kg, a normal maintenance dose of 0.8mg/kg and a maximum of 2mg/kg (up to 90mg). The British National Formulary for Children (BNFC) gives the same advice.

However, the European Medicines Agency recommends a starting dose of 0.8mg/kg per dose which is, therefore, the standard starting dose now. Some patients achieve symptom and biochemical control on less than 0.8 mg/kg per dose. They may be exposed to higher doses than necessary.

To date, approximately 200 patients have started on Burosumab in England. They are all managed by specialist centres. The rare status of XLH means there are relatively few patients in each centre. Treatment effects and trends can only be described by collating data from multiple centres.

The investigators will undertake a review across multiple English centres of the doses of Burosumab. The review will only collect data already in the patients' health records. It will look at factors affecting the starting dose. The investigators will assess the association between dose, blood markers and growth.

DETAILED DESCRIPTION:
X-linked hypophosphatemia (XLH) is a rare, lifelong genetic disorder caused by inactivating mutations in the PHEX gene, leading to elevated levels of fibroblast growth factor 23 (FGF23), which induces renal phosphate wasting. The resultant hypophosphataemia disrupts bone mineralisation, causing rickets, skeletal deformities, growth failure, and chronic pain.

Historically, treatment has relied on oral phosphate and activated vitamin D analogues, which are burdensome and only partially effective. Burosumab (Crysvita), a monoclonal antibody that targets and neutralizes FGF23, is a transformative therapy for XLH. It has been shown to normalise serum phosphate levels, improve growth parameters, and reduce rickets severity. However, real-world data on optimal dosing regimens remain limited.

This study is a multi-centre, pragmatic, retrospective observational analysis conducted across paediatric metabolic bone centres in England. The objective is to assess whether a starting dose of less than 0.8 mg/kg of Burosumab is effective in achieving biochemical control and to characterise dosing variation and outcomes across centres. The current standard dose recommended by the European Medicines Agency (EMA) is 0.8 mg/kg every two weeks, but clinical experience and historical trial data suggest that a proportion of patients may achieve biochemical control on lower doses.

This study will review data from paediatric patients with a diagnosis of XLH who have received at least 12 months of continuous Burosumab treatment under paediatric dosing criteria. Patients will be included regardless of whether they subsequently transitioned to adult dosing, provided their data under paediatric treatment can be clearly delineated.

Data will be extracted from existing clinical records by each participating centre. These records form part of routine care and include biochemistry (serum phosphate, calcium, alkaline phosphatase, creatinine, parathyroid hormone; and urinary calcium, phosphate, and creatinine), auxology (height, weight, sitting height), treatment timelines, imaging findings (notably nephrocalcinosis), and documented adverse effects. Data will be submitted in pseudonymised form through a secure portal hosted by the University of Nottingham.

Data Quality and Registry Procedures:

A data dictionary has been developed to define all collected variables, including normal ranges and units, and to standardise input across sites.

Data validation and consistency checks will be performed at the time of upload, using range and logic rules.

Where needed, study investigators may request clarification or source verification from submitting centres for apparent anomalies or missing data.

All data will be stored on encrypted and access-controlled servers. Backups are performed daily, and all transmissions are encrypted.

Data will be reviewed centrally, and queries raised where missing, inconsistent, or out-of-window data are identified.

A formal statistical analysis plan has been developed. It includes descriptive analyses (means, medians, ranges, and SDs), between-group comparisons using parametric or non-parametric tests as appropriate, and subgroup analyses based on starting dose, PTH status, and age at treatment initiation.

No direct patient contact is involved. Ethical approval will be obtained and, in accordance with UK Health Research Authority guidance and GDPR, individual consent is not required because the study uses fully pseudonymised data collected as part of usual care.

Sample size justification: A minimum of 35 patients started on less than 0.8 mg/kg is required to ensure that the 95% confidence interval for the estimated proportion achieving biochemical control does not cross zero, based on a conservative effect estimate of 10%. Inclusion of additional patients treated at or above 0.8 mg/kg enables robust secondary and comparative analyses.

Missing data strategy: Where values are not available for key time points, interpolation from adjacent data will be used when possible (e.g., to estimate a 6-month height using 3- and 9-month values).

The study is being coordinated by the University of Nottingham and led by Dr James Law Honorary Clinical Associate Professor and Dr Pooja Sachdev, Clinical Associate Professor in Paediatric Endocrinology and Diabetes. Collaborators include national experts in metabolic bone disease. No external funding has been received; centres are contributing data using existing staff and infrastructure.

This study aims to improve understanding of the real-world use of Burosumab and support optimisation of dosing strategies to ensure effective, safe, and cost-conscious care for children with XLH.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of x-linked hypophosphataemia (XLH) including genetic confirmation of a PHEX mutation.
* Has received at least 12 months of continuous Burosumab treatment under paediatric criteria (given Burosumab is not started till a child is 12 months old in England, the minimum age will, therefore, be 2 years old) prior to their 18th birthday.

Exclusion Criteria:

* Burosumab received under adult criteria (patients who have received both Burosumab under paediatric arrangements and, subsequently, adult arrangements, can have data obtained during paediatric dosing included).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with XLH treated with Burosumab under the care of participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved biochemical control (serum phosphate above the lower limit of the local reference range) on a dose of less than 0.8 mg/kg per dose of Burosumab. | During study period, up to 1 year

SECONDARY OUTCOMES:
Comparison of outcomes for patients started on Burosumab at a dose of less than 0.8 mg/kg per dose with those started on a dose of 0.8 mg/kg per dose and above - time to biochemical control | 12 months following first dose of Burosumab
  • Mean difference in time to achieve biochemical control (serum phosphate above the lower limit of the local reference range).
Comparison of outcomes for patients started on Burosumab at a dose of less than 0.8 mg/kg per dose with those started on a dose of 0.8 mg/kg per dose and above - change in height SDS | 12 months following first dose of Burosumab
  • Mean difference in change in height SDS after 12 months of treatment.
Comparison of outcomes for patients started on Burosumab at a dose of less than 0.8 mg/kg per dose with those started on a dose of 0.8 mg/kg per dose and above - dose difference | 12 months following first dose of Burosumab
  • Mean difference in dose of Burosumab at 12 months after first dose.
Comparison of outcomes for patients started on Burosumab at a dose of less than 0.8 mg/kg per dose with those started on a dose of 0.8 mg/kg per dose and above - cost difference | 12 months following first dose of Burosumab
  • Mean difference in cost of giving Burosumab.
Comparison of patients with a raised baseline PTH (prior to initiation of Burosumab) to those with a normal PTH - dose difference | 12 months following first dose of Burosumab
  • Mean difference in dose of Burosumab required to achieve biochemical control (serum phosphate above the lower limit of the local reference range).
Comparison of patients with a raised baseline PTH (prior to initiation of Burosumab) to those with a normal PTH - time to control | 12 months following first dose of Burosumab
  • Mean difference in time to achieve biochemical control.
Comparison of patients with a raised baseline PTH (prior to initiation of Burosumab) to those with a normal PTH - change in height SDS | 12 months following first dose of Burosumab
  • Mean difference in change in height SDS after 12 months of treatment.
Factors influencing dosing regimen in patients on Burosumab | At baseline, first dose of Burosumab
  Analysis using model comparison (additive and subtractive ANOVA models) to assess the association between initial Burosumab dose (mg/kg per dose) and the following patient-related factors:
  1. Calendar year of Burosumab initiation
  2. Age at treatment initiation (years)
  3. Time from diagnosis of XLH to Burosumab initiation (months)
  4. Duration of prior conventional treatment (months)
  Each factor will be included in models predicting Burosumab dose (mg/kg per dose). The relative importance of each predictor will be determined through model fit statistics (e.g., AIC, adjusted R²).
Description of progression and monitoring following the initiation of Burosumab - PTH | From first dose of Burosumab to 12 months later
  • Description of baseline PTH (low, normal, high) and change following treatment (stable, temporary fall, persistent fall, temporary rise, persistent rise).
Description of progression and monitoring following the initiation of Burosumab - nephrocalcinosis | From first dose of Burosumab to 12 months later
  • Proportion of patients with new/deterioration in nephrocalcinosis.
Description of progression and monitoring following the initiation of Burosumab - urinary calcium & phosphate | From first dose of Burosumab to 12 months later
  • Mean change in urinary calcium and phosphate excretion.
Description of progression and monitoring following the initiation of Burosumab - adverse events | From first dose of Burosumab to 12 months later
  • Qualitative description of other reported adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: James Law, BMBS, PhD, MRCPCH, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers may request access to fully anonymised or aggregated summary data by contacting the Chief Investigator. Access will not be granted to case report forms or source documentation.
Supporting Information: Study Protocol
Time Frame: January 2026 for 7 years
Access Criteria: The study protocol will be uploaded to the University of Nottingham Research Data Repository and will be publicly available.
  This study uses pseudonymised clinical data collected as part of routine care from patients with X-linked hypophosphataemia (XLH) across multiple NHS centres. Due to the rarity of XLH and the risk of re-identification, individual participant data (IPD) will not be made publicly available. However, researchers may request access to fully anonymised or aggregated summary data by contacting the Chief Investigator. Requests will be reviewed by the study team and may be granted for appropriate academic or clinical research purposes, subject to a data-sharing agreement and compliance with GDPR and ethical approvals. Access will not be granted to case report forms, or source documentation.

REFERENCES:
- [Background] Saraff V, Nadar R, Hogler W. New Developments in the Treatment of X-Linked Hypophosphataemia: Implications for Clinical Management. Paediatr Drugs. 2020 Apr;22(2):113-121. doi: 10.1007/s40272-020-00381-8. PMID 31965544
- [Background] Padidela R, Cheung MS, Saraff V, Dharmaraj P. Clinical guidelines for burosumab in the treatment of XLH in children and adolescents: British paediatric and adolescent bone group recommendations. Endocr Connect. 2020 Oct;9(10):1051-1056. doi: 10.1530/EC-20-0291. PMID 33112809
- [Background] Imel EA, Glorieux FH, Whyte MP, Munns CF, Ward LM, Nilsson O, Simmons JH, Padidela R, Namba N, Cheong HI, Pitukcheewanont P, Sochett E, Hogler W, Muroya K, Tanaka H, Gottesman GS, Biggin A, Perwad F, Mao M, Chen CY, Skrinar A, San Martin J, Portale AA. Burosumab versus conventional therapy in children with X-linked hypophosphataemia: a randomised, active-controlled, open-label, phase 3 trial. Lancet. 2019 Jun 15;393(10189):2416-2427. doi: 10.1016/S0140-6736(19)30654-3. Epub 2019 May 16. PMID 31104833
- [Background] Carpenter TO, Whyte MP, Imel EA, Boot AM, Hogler W, Linglart A, Padidela R, Van't Hoff W, Mao M, Chen CY, Skrinar A, Kakkis E, San Martin J, Portale AA. Burosumab Therapy in Children with X-Linked Hypophosphatemia. N Engl J Med. 2018 May 24;378(21):1987-1998. doi: 10.1056/NEJMoa1714641. PMID 29791829